CLINICAL TRIAL: NCT00672776
Title: Effects of Paxil CR on Neural Circuits in PTSD
Brief Title: Effects of Paxil CR on Neural Circuits in Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, J. Douglas Bremner, M.D., Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00024970
Record Dates: First submitted 2008-05-01; First posted 2008-05-06 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: hippocampus; paroxetine; stress; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): paroxetine
  Interventions: Drug: paroxetine
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: paroxetine
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
Posttraumatic stress disorder (PTSD) is a major public health problem in this country. It is estimated that at least one out of every seven women in our society have been the victim of childhood sexual abuse at least once before their 18th birthday. Previous studies have shown that stress is associated with damage to neurons of the hippocampus, a brain area involved in learning and memory. Also, imaging studies of brain function are consistent with dysfunction of the medial prefrontal cortex during presentation of traumatic cues. We have previously shown that serotonin reuptake inhibitor medications (paroxetine; Paxil) can change memory function and hippocampal structure in PTSD. We now propose to perform a placebo controlled study with Paxil CR (paroxetine hydrochloride controlled-release tablets), which is thought as paroxetine with less side-effects. The main purpose of this study is to determine the effects of Paxil CR on memory deficits measured with neuropsychological testing, hippocampal volume measured with a magnetic resonance imaging (MRI), medial prefrontal lobe cortical function estimated with PET, and cortisol response (reflecting the intensity of stress) in men and women with PTSD. We plan to recruit 40 subjects. After completing physical examination and evaluating neuropsychiatric history, patients will undergo an initial group of tests which includes memory testing, MRI and PET brain scan, and measurement of cortisol in their saliva. Afterwards, half will receive Paxil CR 12.5 to 62.5 mg and half will receive a placebo (sugar pill) in the beginning of the first 12 weeks as "Double Blind Phase". After 12 weeks, they will be administered memory tests, PET and MRI scan for the post-treatment phase. After this period, Paxil CR will be offered to the placebo group and followed for an additional 12 weeks. They will have final memory tests, and a MRI scan. We hypothesize that Paxil CR exerts its efficacy by acting on abnormal neural circuits, including hippocampus and prefrontal cortex, in PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients meeting Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV) criteria for PTSD assessed by the Structured Clinical Interview for DSM IV (SCID).
* All patients with PTSD will be greater than 18 years of age, and will be required to give informed consent.
* Patients will be recruited from newspaper advertisements and fliers.
* All patients must be free of major medical illness on the basis of history and physical examination, lab testing, and electrocardiogram, and must not be actively abusing substances or alcohol.
* Patients should be free of psychotropic medications for four weeks before the study.

Exclusion Criteria:

* Pregnant and breast-feeding women will not be studied. Female subjects will be required to have a negative pregnancy test before the study. Female subjects of childbearing age will be advised to use barrier contraception for the duration of the study, in addition to other forms of contraception that they may be using.
* Serious medical or neurological illness or a hypersensitivity to paroxetine.
* Past or present steroid use.
* Electroconvulsive therapy (ECT) within the 6 months prior to study entry.
* Organic mental disorders or epilepsy
* History of head trauma
* Cerebral infectious disease or dyslexia.
* History of psychosis, schizophrenia, or eating disorders.
* Active suicidality or homicidality

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2003-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Brain Function with Traumatic Reminders | three months
  PET measurement of brain activation before and after paroxetine or placebo treatment.